CLINICAL TRIAL: NCT00721422
Title: A Phase 1, Open-Label, Single Dose Study To Evaluate The Pharmacokinetics, Safety, And Tolerability Of PD 0332334 In Subjects With Various Degrees Of Renal Function
Brief Title: A Single Dose Study Investigating the Elimination as Well as the Tolerability of PD 0332334 in Healthy Subjects as Compared to Patients With Impaired Kidney Function.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Please see Detailed Description for termination reason.
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: A5361023
Record Dates: First submitted 2008-07-22; First posted 2008-07-24 (Estimated); Last update posted 2010-02-17 (Estimated); Status verified 2010-02

CONDITIONS: Renal Insufficiency; Pharmacokinetics
Keywords: Pharmacokinetics of PD 0332334 in subjects with renal insufficiency
MeSH Terms: conditions — Renal Insufficiency | interventions — imagabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1-Normal (Experimental)
  Interventions: Drug: PD 0332334
- Group 2-Mild (Experimental)
  Interventions: Drug: PD 0332334
- Group 3-Moderate (Experimental)
  Interventions: Drug: PD 0332334
- Group 4-Severe (Experimental)
  Interventions: Drug: PD 0332334

INTERVENTIONS:
Drug: PD 0332334 — 50 mg (two 25 mg capsules), single, oral dose
  Other Names: imagabalin
  Arms: Group 1-Normal
Drug: PD 0332334 — 50 mg (two 25 mg capsules), single, oral dose
  Arms: Group 2-Mild
Drug: PD 0332334 — 50 mg (two 25 mg capsules), single, oral dose
  Arms: Group 3-Moderate
Drug: PD 0332334 — 50 mg (two 25 mg capsules), single, oral dose
  Arms: Group 4-Severe

SUMMARY:
1. To investigate the effect of kidney function on the elimination of a single dose of PD 0332334 from the body.
2. To investigate the safety and tolerability of a single dose of PD 0332334 in patients with impaired kidney function.

DETAILED DESCRIPTION:
Additional Study Purpose Details: Investigation of the pharmacokinetics, safety, and tolerability of a single dose of PD 0332334 in patients with impaired renal function.

On February 23rd 2009, a decision to terminate further development for PD 0332334 was communicated to investigators in this study. The decision to terminate this study was not based on any safety concerns.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers OR subjects with kidney impairment

Exclusion Criteria:

1. Receiving hemodialysis
2. clinically significant or unstable medical disease other than kidney disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-08; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
maximum plasma concentration (Cmax), time of maximum plasma concentration (Tmax), and apparent clearance from plasma (CL/F) | 1 day
amount of PD 0332334 eliminated unchanged in urine during the 96-hour collection period (Ae96) | 5 days
PD 0332334 area under the curve from 0 to infinity (AUCinf), PD 0332334 area under the curve from 0 to last quantifiable concentration (AUClast), | 5 to 17 days depending on cohort
PD 0332334 renal clearance (CLr), apparent volume of distribution (Vz/F), terminal half life (t1/2), | 5 to 17 days depending on cohort

SECONDARY OUTCOMES:
Adverse events, ECG, physical exams, clinical safety laboratory, and vital signs | 5 to 17 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Pfizer Investigational Site, Cypress, California
  - Pfizer Investigational Site, Miami, Florida

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5361023&StudyName=A%20single%20dose%20study%20investigating%20the%20elimination%20as%20well%20as%20the%20tolerability%20of%20PD%200332334%20in%20healthy%20subjects%20as%20compared%20to%20patie